CLINICAL TRIAL: NCT05665647
Title: An Open Labe Study to Evaluate the Drug-Drug Interaction of Itraconazole, Rifampicin and Midazolam With SIM0417/Ritonavir in Healthy Adult Chinese Participants
Brief Title: Drug-Drug Interaction Study of Itraconazole, Rifampicin and Midazolam With SIM0417/Ritonavir in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIM0417-107
Record Dates: First submitted 2022-12-19; First posted 2022-12-27 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: Drug-drug interaction
MeSH Terms: interventions — Ritonavir; Itraconazole; Rifampin; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: SIM0417/ritonavir and itraconazole (Experimental): Interaction between SIM0417/ritonavir and itraconazole
  Interventions: Drug: Cohort 1: SIM0417/ritonavir and itraconazole
- Cohort 2: SIM0417/ritonavir and rifampicin (Experimental): Interaction between SIM0417/ritonavir and rifampicin
  Interventions: Drug: Cohort 2: SIM0417/ritonavir and rifampicin
- Cohort 3: SIM0417/ritonavir and midazolam (Experimental): Interaction between SIM0417/ritonavir and midazolam
  Interventions: Drug: Cohort 3: SIM0417/ritonavir and midazolam

INTERVENTIONS:
Drug: Cohort 1: SIM0417/ritonavir and itraconazole — SIM0417/Ritonavir: Dose: 750 mg SIM0417 coadministered with 100 mg ritonavir once: Day1-Day2, Day9-Day10, BID; Day3,Day11(once only in the morning); Itraconazole：Dose: 200mg once；Day6-Day13, QD
  Other Names: Interaction between SIM0417/ritonavir and itraconazole
  Arms: Cohort 1: SIM0417/ritonavir and itraconazole
Drug: Cohort 2: SIM0417/ritonavir and rifampicin — SIM0417/Ritonavir:Dose: 750 mg SIM0417 coadministered with 100 mg ritonavir once: Day1,Day11(once only in the morning); Rifampicin：Dose: 0.6g once; Day4-Day12, QD
  Other Names: Interaction between SIM0417/ritonavir and rifampicin
  Arms: Cohort 2: SIM0417/ritonavir and rifampicin
Drug: Cohort 3: SIM0417/ritonavir and midazolam — SIM0417/Ritonavir: 750 mg SIM0417 coadministered with 100 mg ritonavir, Day3-Day6, BID; Day7(once only in the morning) Midazolam：Dose: 2mg once; Day1, Day6, QD
  Other Names: Interaction between SIM0417/ritonavir and midazolam
  Arms: Cohort 3: SIM0417/ritonavir and midazolam

SUMMARY:
This is a phase 1, open-label, fixed-sequence, 2-period drug-drug interaction study to evaluate the pharmacokinetic interactions of itraconazole, rifampicin, midazolam, and SIM0417/ritonavir in healthy Chinese subjects.

DETAILED DESCRIPTION:
This is a phase 1, open-label, fixed-sequence, 2-period drug-drug interaction study which was divided into three cohorts.

Cohort 1: to evaluate the effect of the CYP3A4 inhibitor itraconazole on the pharmacokinetics of SIM0417 and ritonavir in healthy participants.

Cohort 2: to evaluate the effect of the CYP3A4 inducer rifampicin on the pharmacokinetics of SIM0417 and ritonavir in healthy participants.

Cohort 3: to evaluate the effect of SIM0417/ ritonavir on the pharmacokinetics of CYP3A4 substrate midazolam in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the research content, process, and potential risks of this trial, voluntarily participate in the clinical trial and sign the informed consent,
2. Healthy male and female subjects aged ≥18 years and ≤45 years old.
3. Male weight ≥50kg, female weight ≥45kg, body mass index ≥19 kg/m2 and ≤28 kg/m2.
4. Subjects agree to use generally accepted effective contraception from the time they sign the informed consent form. And female subjects of Cohort 1 agree to take recognized effective contraceptive measures during the study period and for the next menstrual cycle after the last dose of the study drug (male subjects up to 1 month after the last dose of the study drug ). Subjects of cohort 2 agree to take recognized effective contraceptive measures during the study period and within 1 month after the last dose of the study drug. Subjects of cohort 3 agree to take recognized effective contraceptive measures during the study period and within 3 months after the last dose of the study drug. Female subjects had been using effective contraception for 14 days prior to screening.

Exclusion Criteria:

1. Any diseases that may affect the study results or the safety and status of the subjects, including but not limited to the central nervous system, respiratory system, cardiovascular system, alimentary system, blood and lymphatic system, endocrine system, musculoskeletal system, hepatic and kidney function obstacle.
2. Difficulty in venous blood collection, a history of fainting blood or needles, or those who cannot tolerate blood collection with intravenous indwelling needles.
3. With dysphagia or any history of gastrointestinal diseases that affect drug absorption.
4. Have special requirements for diet and cannot comply with the diet provided and corresponding regulations.
5. With specific allergic history ( asthma, urticaria, eczema, etc. ) or allergic constitution ( such as those allergic to two or more drugs, food such as milk, and pollen ) or allergic to any component of the research drug or research drug.
6. With special diet ( including pitaya, mango, grapefruit, food or beverage containing caffeine, etc. ) or intense exercise taken within 48 h before the first administration of the drug.
7. Taken of any prescription, non-prescription, vitamin, or herbal medicine within 4 weeks before and during the screening period and/or any vitamin, health care products were taken within 2 weeks before and during the screening period.
8. During the first 3 months prior to screening or from the screening period to the first administration period, alcohol was often consumed, i.e., more than 2 units of alcohol per day ( 1 unit = 360 mL beer or 45 mL spirits with 40 % alcohol or 150 mL wine ); or alcohol breath test positive.
9. More than 5 cigarettes per day during the 3 months prior to screening.
10. Participated in any drug clinical trial as a subject within 3 months prior to screening and took the study drug.
11. With blood donation or blood loss greater than 200 mL within 3 months prior to screening, or blood transfusion or blood products were received within 4 weeks.
12. Have a history of drug abuse or a positive drug abuse screen.
13. At the time of screening or baseline, the blood pressure in the resting state and the pulse are within the following ranges: such as systolic blood pressure <90 mmHg or ≥140 mmHg, diastolic blood pressure <60 mmHg or ≥90 mmHg, pulse <55 bpm or >100 bpm.
14. Electrocardiographic QTc > 450 msec (Fridericia formula) at screening and/or baseline, or presence of risk factors for Torsade de Pointes (eg, history of heart failure, history of hypokalemia, family with prolonged QT syndrome) history), or other abnormal clinical significance (judged by the investigator).
15. HBV surface antigen, HCV antibody, HIV, or syphilis are positive during screening.
16. Physical examination, vital signs, ECG, blood routine, blood biochemistry ( serum creatinine, total bilirubin> 1.0 × ULN, ALT, AST, triglyceride>1.1 ULN)), coagulation function, thyroid function, urine routine, chest X-ray, abdominal B-scan ultrasonography results were abnormal and have clinical significance (judged by the investigator).
17. Those who have been vaccinated within 1 month before screening, or have been vaccinated with a COVID-19 vaccine within 1 week before screening, or plan to be vaccinated during the treatment or within 2 weeks after the last dose of study drug.
18. Be positive in SARS-CoV-2 nucleic acid test at screening.
19. Those who had undergone major surgery within 6 months prior to screening or were scheduled to undergo surgery during the study period and were determined by the investigators to be unsuitable for inclusion.
20. Subjects have acute disease with clinical significance that judged unsuitable for inclusion judged by the investigator within 1 month before screening.
21. Females who are pregnant or breastfeeding or positive result from pregnancy test.
22. Subjects have other conditions that are not suitable for participating in this research, or the subjects may not be able to complete this research for other reasons (judged by the investigator).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-02-14 (Actual)

PRIMARY OUTCOMES:
Cmax of SIM0417 in cohort 1 | Up to Day 14
  Cmax of SIM0417 when SIM0417/ritonavir is multiple administered or combined with itraconazole
Ctrough of SIM0417 in cohort 1 | Up to Day 14
  Ctrough of SIM0417 when SIM0417/ritonavir is multiple administered or combined with itraconazole
AUC0-t of SIM0417 in cohort 1 | Up to Day 14
  AUC0-t of SIM0417 when SIM0417/ritonavir is multiple administered or combined with itraconazole
AUC0-∞ of SIM0417 in cohort 1 | Up to Day 14
  AUC0-∞ of SIM0417 when SIM0417/ritonavir is multiple administered or combined with itraconazole
AUCtau of SIM0417 in cohort 1 | Up to Day 14
  AUCtau of SIM0417 when SIM0417/ritonavir is multiple administered or combined with itraconazole
t1/2 of SIM0417 in cohort 1 | Up to Day 14
  t1/2 of SIM0417 when SIM0417/ritonavir is multiple administered or combined with itraconazole
Cmax of SIM0417 in cohort 2 | Up to Day 14
  Cmax of SIM0417 when SIM0417/ritonavir is single dosed administration or combined with rifampicin
AUC0-t of SIM0417 in cohort 2 | Up to Day 14
  AUC0-t of SIM0417 when SIM0417/ritonavir is single dosed administration or combined with rifampicin
AUC0-∞ of SIM0417 in cohort 2 | Up to Day 14
  AUC0-∞ of SIM0417 when SIM0417/ritonavir is single dosed administration or combined with rifampicin
t1/2 of SIM0417 in cohort 2 | Up to Day 14
  t1/2 of SIM0417 when SIM0417/ritonavir is single dosed administration or combined with rifampicin
Cmax of midazolam | Up to Day 9
  Cmax of midazolam when midazolam is single dosed administration or combined with SIM0417/ritonavir
AUC0-t of midazolam | Up to Day 9
  AUC0-t of midazolam when midazolam is single dosed administration or combined with SIM0417/ritonavir
AUC0-∞ of midazolam | Up to Day 9
  AUC0-∞ of midazolam when midazolam is single dosed administration or combined with SIM0417/ritonavir
t1/2 of midazolam | Up to Day 9
  t1/2 of midazolam when midazolam is single dosed administration or combined with SIM0417/ritonavir

SECONDARY OUTCOMES:
Adverse Events of Cohort 1 | Up to Day 26
  Number of Participants With Adverse Events
Adverse Events of Cohort 2 | Up to Day 25
  Number of Participants With Adverse Events
Adverse Events of Cohort 3 | Up to Day 20
  Number of Participants With Adverse Events
Vital Signs | Up to Day 14
  Number of Participants With Clinically Notable Vital Signs
ECG | Up to Day 14
  Number of Participants With Clinically Notable Electrocardiogram (ECG) Values
Laboratory Tests | Up to Day 14
  Number of Participants With Clinically Notable Laboratory Tests
Cmax of ritonavir in Cohort 1 | Up to Day 14
  Cmax of ritonavir when SIM0417/ritonavir is multiple administered or combined with itraconazole
Ctrough of ritonavir in Cohort 1 | Up to Day 14
  Ctrough of ritonavir when SIM0417/ritonavir is multiple administered or combined with itraconazole
AUC0-t of ritonavir in Cohort 1 | Up to Day 14
  AUC0-t of ritonavir when SIM0417/ritonavir is multiple administered or combined with itraconazole
AUC0-∞ of ritonavir in Cohort 1 | Up to Day 14
  AUC0-∞ of ritonavir when SIM0417/ritonavir is multiple administered or combined with itraconazole
AUCtau of ritonavir in Cohort 1 | Up to Day 14
  AUCtau of ritonavir when SIM0417/ritonavir is multiple administered or combined with itraconazole
t1/2 of ritonavir in Cohort 1 | Up to Day 14
  t1/2 of ritonavir when SIM0417/ritonavir is multiple administered or combined with itraconazole
Cmax of ritonavir in Cohort 2 | Up to Day 14
  Cmax of ritonavir when SIM0417/ritonavir is single dosed administration or combined with rifampicin
AUC0-t of ritonavir in Cohort 2 | Up to Day 14
  AUC0-t of ritonavir when SIM0417/ritonavir is single dosed administration or combined with rifampicin
AUC0-∞ of ritonavir in Cohort 2 | Up to Day 14
  AUC0-∞ of ritonavir when SIM0417/ritonavir is single dosed administration or combined with rifampicin
t1/2 of ritonavir in Cohort 2 | Up to Day 14
  t1/2 of ritonavir when SIM0417/ritonavir is single dosed administration or combined with rifampicin

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Principal Investigator — Shandong First Medical University
Locations (1):
- Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ye PP, Yao BF, Yang Y, Yang XM, Li Q, Song LL, Chen KG, Zhou HY, Shi JY, Zhang YH, Zhao FR, Guo ZJ, Xu SS, Chen J, Goh AH, Zhu SW, Zheng Y, Zhao W. Drug-drug interactions of simnotrelvir/ritonavir: an open-label, fixed-sequence, two-period clinical trial. Clin Microbiol Infect. 2025 Jan;31(1):101-107. doi: 10.1016/j.cmi.2024.09.007. Epub 2024 Sep 18. PMID 39299559